CLINICAL TRIAL: NCT07213843
Title: Combined Circulatory and Dietary Interventions for Neuropathy (CDIN)
Brief Title: Combined Circulatory and Dietary Interventions for Neuropathy
Acronym: CDIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Kyan Sahba, Principal Invetigator, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5250381
Record Dates: First submitted 2025-09-25; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Diabete Type 2; Neuropathy, Painful
Keywords: neuropathy; diabetes type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Neuropathy, Painful

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel assignment study with three active treatment arms (INF® therapy only, NVIf only, and INF® + NVIf) to compare their effects on neuropathy symptoms
Masking Description: This study uses an open-label design with no masking; both participants and study personnel will know the assigned treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- INF® Therapy Only Group (Experimental): INF® therapy is a manual technique designed to improve neural circulation by using a series of manual holds administered by a trained practitioner. Participants will receive 60-minute sessions, 2-3 times per week, for a total of 8 sessions.
  Interventions: Other: INF® Therapy
- NVIf Only Group (Experimental): NVIf, is a dietary intervention that uses a patented ultrasound technology to assess vascular responses to food allergens. By identifying foods that exacerbate inflammation and restrict circulation, the intervention guides patients to eliminate these foods, thereby improving nerve health. Those in this group will participate in follow-up for food elimination adherence, including daily tracking of foods ingested. Week 1-2: 4 x NVI food guided-elimination visits. Week 2-5 complete weekly Likert scale inquiring about food eliminations and weekly phone call check-in attempts will be made by research staff.
  Interventions: Other: NVIf
- INF® Therapy + NVIf Group (Experimental): INF® therapy and NVI Food-Guided Elimination Group: Week 1-2: 4 x NVI food guided-elimination visits. Participants will receive 60-minute sessions, 2-3 times per week, for a total of 8 sessions. As well as participate in NVIf, which is a dietary intervention that uses a patented ultrasound technology to assess vascular responses to food allergens. By identifying foods that exacerbate inflammation and restrict circulation, the intervention guides patients to eliminate these foods, thereby improving nerve health. Those in this group will participate in follow-up for food elimination adherence, including daily tracking of foods ingested. Week 2-5 complete weekly Likert scale inquiring about food eliminations and weekly phone call check-in attempts will be made by research staff as well as INF® therapy for 60-minute sessions, 2-3 times per week, for a total of 8 sessions.
  Interventions: Other: INF® Therapy; Other: NVIf

INTERVENTIONS:
Other: INF® Therapy — INF® therapy is a manual technique designed to improve neural circulation by using a series of manual holds administered by a trained practitioner,
  Other Names: Intranerual Facilitation
  Arms: INF® Therapy + NVIf Group; INF® Therapy Only Group
Other: NVIf — NVIf is a dietary intervention that uses a patented ultrasound technology to assess vascular responses to food allergens
  Other Names: Neuro vascular index food-guided elimination
  Arms: INF® Therapy + NVIf Group; NVIf Only Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of three different interventions in improving neuropathy symptoms in individuals aged 35-85 with moderate to severe neuropathy. The study will compare three treatment groups: Intraneural Facilitation® (INF®) therapy alone, INF® therapy combined with Neuro vascular index (NVI) food-guided elimination (NVIf), and NVIf alone. The aim is to determine which treatment results in the greatest improvement in neuropathy symptoms, including quality of life, sensory and pain improvements, and functional outcomes.

DETAILED DESCRIPTION:
The purpose of this investigator-initiated study is to observe the effectiveness of a manual physical therapy technique known as Intraneural Facilitation (INF®), both independently and in combination with a Nutritional Vascular Inflammation focused (NVIf) dietary intervention, in improving neurovascular function, pain, and physical performance in individuals with moderate to severe peripheral neuropathy (PN). Subjects will be randomized into one of the three interventions arms: (1) INF® therapy alone, (2) NVIf intervention alone or (3) a combination of both. INF® is a manual therapy, while NVIf utilizes ultrasound guided food elimination. Outcomes include pain (Visual analog scale), sensory function (Semmes Weinstein Monofilament), physical function (Lower extremity functional scale, 10-meter walk test, timed up and go) quality of life (Norfolk Quality of life-Diabetic neuropathy), and neurovascular blood flow analysis. Study participants will be 35-85 years old with a physician-confirmed diagnosis of moderate to severe lower extremity peripheral neuropathy and at least one symptom: numbness, tingling, burning, sharp pain, or increased sensitivity. They must score 0-60 on the Lower Extremity Functional Scale (LEFS), speak and understand English, provide written informed consent, and be willing to complete all study procedures, including intervention and follow-up visits. Participants must be able to ambulate independently with or without an assistive device. Subjects will be recruited using email and flyer through the Neuropathic Therapy Center (NTC) research interest list and through providers at Loma Linda's University (LLU) Health offices. 60 subjects will be recruited, and consent will take place at the LLU or at the Murrieta study site prior to randomization, administered by trained study staff authorized to obtain informed consent.

ELIGIBILITY:
Inclusion Criteria

* Confirmed diagnosis of peripheral neuropathy in the lower extremities by a physician
* Lower Extremity Functional Scale (LEFS) score between 0-60 (indicating moderate to significant difficulty in lower extremity function)
* Ability to speak and understand English
* Ability to provide appropriate written informed consent
* Willingness to participate in all study procedures, including the intervention and follow-up visits
* Ability to ambulate independently with or without an assistive device

Exclusion Criteria

* Any medical condition suggesting potential decline in function over the next 6 months (e.g., ongoing chemotherapy, radiation therapy, or dialysis)
* Active alcohol or drug misuse
* End-stage renal failure
* Uncontrolled hypertension
* Severe dyslipidemia
* Chronic liver disease
* Autoimmune disease
* Advanced chronic obstructive pulmonary disease (COPD)
* Active inflammation
* Shingles-related neuropathy
* Presence of any lower extremity amputations or significant wounds
* Severe chronic medical conditions requiring active treatment that could interfere with study outcomes
* Morbid obesity
* Concomitant use of medications or devices that may interfere with study results or are not allowed per protocol
* Inability to comprehend or provide informed consent
* Inability to speak or understand English
* Pregnancy, breastfeeding, or planning pregnancy during the study period (female participants)
* Inability or unwillingness to adhere to study procedures, including dietary guidelines or follow-up visits
* Inability to complete all required study assessments, including follow-up appointments and questionnaires

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity | Baseline (Week 0) and post-intervention (Week 4-5)
  Pain intensity will be assessed using the Visual Analog Scale. Improvement will be indicated by reduced VAS scores. Unit of Measure: Millimeters on a 0-100 mm scale.
Change in Sensory Function | Baseline (Week 0), mid-treatment (Week 3), and post-intervention (Week 4-5)
  Sensory function will be assessed using the Semmes-Weinstein Monofilament test. Improvement will be indicated by increased monofilament detection. Detection threshold in grams (monofilament response: detected/not detected)
Change in Functional Limitation | Baseline (Week 0) and post-intervention (Week 4-5)
  Functional limitation related to neuropathy will be assessed using the Lower Extremity Functional Scale. Improvement will be indicated by higher Lower Extremity Functional Scale scores. Scale score (0-80).
Change in Gait Speed | Baseline (Week 0), mid-treatment (Week 3), and post-intervention (Week 4-5)
  Gait speed will be assessed using the 10-Meter Walk Test. Improvement will be indicated by faster walk time. Seconds to complete 10 meters (converted to meters/second if applicable)
Change in Mobility and Fall Risk | Baseline (Week 0), mid-treatment (Week 3), and post-intervention (Week 4-5)
  Mobility and fall risk will be assessed using the Timed Up and Go (TUG) test. Improvement will be indicated by shorter completion times. Unit of Measure: Seconds.

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline (Week 0) and post-intervention (Week 4-5)
  Quality of life will be measured using the Norfolk Quality of Life-Diabetic Neuropathy questionnaire to determine the effect of each treatment approach on overall patient well-being. Higher scores indicate greater impairment; a reduction reflects improved quality of life. Lowest score=0, means best quality of life with little to no neuropathy impacts. A maximum score of 138, means worst quality of life with severe impairments.

OTHER OUTCOMES:
Change in Neurovascular Function and Inflammation | Baseline (Week 0) and post-intervention (Week 4-5)
  Mechanistic analysis will be performed using the Neurovascular Index with Philips Affinity 50 Ultrasound to evaluate changes in microvascular resistance and neurovascular blood flow, as well as the effect of NVI-guided food elimination on reducing neurovascular inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Kyan Sahba, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Neuropathic Therapy Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD). De-identified aggregate data may be made available upon reasonable request to the Principal Investigator, following study completion and publication of primary results, in accordance with institutional policies and IRB approval.

REFERENCES:
- See also: A Retrospective Assessment of Neuropathic Pain in Response to Intraneural Facilitation® Therapy and Neurovascular Index-Guided Food Elimination — https://pubmed.ncbi.nlm.nih.gov/40149665/
- See also: Treating peripheral neuropathy in individuals with type 2 diabetes mellitus with intraneural facilitation: a single blind randomized control trial — https://pubmed.ncbi.nlm.nih.gov/35922961/